CLINICAL TRIAL: NCT00720226
Title: Efficacy of Losartan in Preventing Progression of COPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Robert A. Wise, Professor of Medicine (Pulmonary and Critical Care), Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1P50HL084945 (NIH); 1P50HL084945 (NIH); NCT00720044 (obsolete NCT alias)
Record Dates: First submitted 2008-07-18; First posted 2008-07-22 (Estimated); Results first posted 2017-04-25 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-03

CONDITIONS: COPD; Emphysema; Chronic Bronchitis; Smoking
Keywords: COPD; emphysema; angiotensin receptor blocker
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema; Bronchitis, Chronic; Smoking | interventions — Losartan; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Losartan (Experimental): Losartan 100 mg daily
  Interventions: Drug: Losartan
- Placebo (Placebo Comparator): Placebo 1 pill daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Losartan — Losartan 100 mg daily
  Other Names: Cozaar
  Arms: Losartan
Drug: Placebo — Placebo pill daily
  Other Names: "Sugar pill"
  Arms: Placebo

SUMMARY:
Evidence in animals shows that losartan can prevent or reverse inflammation and lung damage due to smoking. The goal of this study is to determine whether this drug which is also used to treat hypertension can stabilize or improve lung function in people who have from chronic obstructive pulmonary disease (COPD).

DETAILED DESCRIPTION:
Participants will be given either losartan in a dose of 50-100 mg per day for a period of one year. During that time, they will have lung function tests, breathing tests, and computed tomograms of the chest. These tests will determine whether there is inflammation in the lung and whether there is progressive involvement of the lung with COPD.

ELIGIBILITY:
Inclusion Criteria:

* Adults with COPD who are either active or former smokers

Exclusion Criteria:

* Clinical requirement or history of intolerance of angiotensin receptor blockers, serious heart, liver, kidney, neurological disease.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2008-07; Primary Completion 2014-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert A. Wise, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Asthma and Allergy Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Limited dataset available to qualified investigators with data use agreement.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Losartan | Placebo
Started | 54 | 52
Completed | 47 (Participants not completing did not have 12 month CT scan) | 48 (Participants not completing did not have 12 month CT scan)
Not Completed | 7 | 4
Not completed — Withdrawal by Subject | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo 1 tablet daily
- Total: Total of all reporting groups
Arm/Group | Losartan | Placebo | Total
Number analyzed (Participants) | 54 | 52 | 106
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.3 (10.0) | 59.3 (9.8) | 58.8 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 25 | 53
  Male | 26 | 27 | 53
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 14 | 30
  White | 38 | 38 | 76
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
FEV1 (L) [Mean (Standard Deviation); unit: L (BTPS)] — Population: Participants with analyzable data pre-bronchodilator
  L (BTPS)
    number analyzed (Participants) | 51 | 51 | 102
    (all) | 1.57 (0.52) | 1.42 (.46) | 1.49 (0.69)
FEV1/FVC (%) [Mean (Standard Deviation); unit: percent] — Ratio of Forced Expiratory Volume in 1 second (FEV1) divided by Forced Vital Capacity (FVC) and then multiplied by 100 to give the ratio in percent. Population: Participants with analyzable data from pre-bronchodilator spirometry
  percent
    number analyzed (Participants) | 51 | 51 | 102
    (all) | 52.9 (10.5) | 49.9 (11.3) | 51.4 (15.4)
Smoking Status [Number; unit: participants]
  Current Smoker | 36 | 36 | 72
  Former Smoker | 18 | 16 | 34
Emphysema on HRCT [Count of Participants; unit: Participants] — Emphysema was measured as percent of lung voxels with Hounsfield units (HU) less than -950 HU. Participants with 5-35% of lung parenchyma with HU < -950 were considered to have radiographic emphysema.
  Participants | 24 | 21 | 45

OUTCOME MEASURES:

1. Primary Outcome: Change in Percent Emphysema on CT Scan
Description: Percent emphysema calculated as percent of CT voxels less than -950 HU measured at TLC. Analysis limited to patients with 5-35% emphysema on CT scan at baseline.
Time Frame: Change between baseline and month 12.
Population: Participants with 5-35% emphysema on baseline CT scan
Measure: Mean (Standard Deviation); unit: % Emphysema Whole Lung
Groups:
- Losartan: Losartan: Losartan 100 mg daily (participants with 5-35% emphysema)
- Placebo: Placebo: Placebo pill daily (Participants with 5-35% emphysema)
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 23 | 20
% Emphysema Whole Lung | -0.32 (3.7) | 2.18 (4.9)
Statistical Analysis 1: Comparison: Losartan vs Placebo; Participants demonstrating 5-35% emphysema on baseline CT scan; Test type: Superiority; p = 0.06, t-test, 2 sided

2. Secondary Outcome: Change in FEV1 (L)
Description: Change in FEV1 (L) post-bronchodilator from baseline to 12 months. Analysis includes only participants with 5-35% emphysema at baseline.
Time Frame: Measured at Baseline and Month 12
Population: Participants with 5-35% emphysema at baseline who had HRCT scans performed both at baseline and at 12 months.
Measure: Mean (Standard Deviation); unit: L (BTPS)
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 23 | 20
L (BTPS) | -0.0879 (0.163) | -0.0581 (0.167)
Statistical Analysis 1: Comparison: Losartan vs Placebo; Participants with 5-35% emphysema at baseline; Test type: Superiority; p = 0.55, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Losartan 100 mg Daily: Losartan 100 mg daily
  Losartan: Losartan 100 mg daily
Arm/Group | Losartan 100 mg Daily | Placebo
All-Cause Mortality (participants affected / at risk) | 0/54 | 1/52
Serious Adverse Events (participants affected / at risk) | 7/54 | 18/52
Other Adverse Events (participants affected / at risk) | 19/54 | 24/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Losartan 100 mg Daily (N=54) | Placebo (N=52)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 18 (18)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Losartan 100 mg Daily (N=54) | Placebo (N=52)
Worsening of respiratory symptoms (Respiratory, thoracic and mediastinal disorders) | 19 (19) | 24 (24)
Worsening of gastrointestinal symptoms (Gastrointestinal disorders) | 7 (7) | 11 (11)
Worsening of musculoskeletal symptoms or fracture (Musculoskeletal and connective tissue disorders) | 8 (8) | 3 (3)

LIMITATIONS AND CAVEATS:
Study was designed as feasibility study for assessment of variability of outcomes and tolerability of treatment in patients with pre-existing emphysema in association with COPD.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No